CLINICAL TRIAL: NCT05499845
Title: Comparison of the Effects of TIVA and Inhalation Anesthesia Methods on Olfactory Functions and Olfactory Memory
Brief Title: Effects of Different Anesthesia on Odor Memory
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2013/02
Record Dates: First submitted 2022-06-02; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Smell Functions; Odor Memory
Keywords: General anesthesia management; propofol; sevoflurane; odor memory; smell functions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group P (n=40) (Propofol),
  Interventions: Diagnostic Test: butanol threshold test and smell identification tests
- Group PS (n=40) (Propofol-Sevoflurane),
  Interventions: Diagnostic Test: butanol threshold test and smell identification tests
- Group S (n=40) (Sevoflurane).
  Interventions: Diagnostic Test: butanol threshold test and smell identification tests

INTERVENTIONS:
Diagnostic Test: butanol threshold test and smell identification tests — no additional intervention

SUMMARY:
This study aimed to research the effect of different general anesthesia administration on postoperative smell functions and memory.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II risk groups
* operated under elective conditions with general anesthesia requiring intubation
* operation durations of 40-180 minutes.

Exclusion Criteria:

* intracranial,
* endocrine or nasal surgery,
* pregnant cases,
* those with history of respiratory tract diseases and psychiatric disease, with disorder of odor reception and perception,
* with smoking and chronic alcohol use,
* requiring a nasogastric probe

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 97
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Butanol Threshold Test | during 24 hour after surgery
  threshold detection and odor discrimination
Odor Identification Test | during 24 hour after surgery
  odor discrimination

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No